CLINICAL TRIAL: NCT06994468
Title: Effect of B-cell Depleting Therapies on PLA2R-specific B Cells in Patients With Membranous Nephropathy
Acronym: DEEPER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DEEPER
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Membranous Nephropathy
Keywords: primary membranous nephropathy; PLA2R-specific B cells; Obinutuzumab; Felzartamab
MeSH Terms: conditions — Glomerulonephritis, Membranous

STUDY DESIGN:
Intervention Model Description: PBMCs will be isolated form both anti-PLA2 positive and anti-PLAR2 negative patients enrolled in the ORION and MONET studies. The anti-PLAR2 negative patients will be sued as negative control patients. In addition, PBMCs will be isolated from volunteers. These PBMCs will serve to set a reference range for the planned analyses, ensuring the absence of confounding factors related to underlying health conditions or pharmacological interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- PBMCs from ORION patients positive for anti-PLAR2 (Experimental): Peripheral Blood Mononuclear Cells (PBMCs) samples identified among anti-PLAR2 positive patients enrolled in the ORION study, who provided consent to store their samples collected during the follow-up at the Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica (BG).
  Interventions: Diagnostic Test: Flow-cytometry tetramer-based antigen-bait assay
- PBMCs from MONET patients positive for anti-PLAR2 (Experimental): Peripheral Blood Mononuclear Cells (PBMCs) samples identified among anti-PLAR2 positive patients enrolled in the MONET study, who provided consent to store their samples collected during the follow-up at the Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica (BG).
  Interventions: Diagnostic Test: Flow-cytometry tetramer-based antigen-bait assay
- PBMCs from ORION patients negative for anti-PLAR2 (Active Comparator): Peripheral Blood Mononuclear Cells (PBMCs) samples identified among anti-PLAR2 negative patients enrolled in the ORION study, who provided consent to store their samples collected during the follow-up at the Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica (BG).
  Interventions: Diagnostic Test: Flow-cytometry tetramer-based antigen-bait assay
- PBMCs from MONET patients negative for anti-PLAR2 (Active Comparator): Peripheral Blood Mononuclear Cells (PBMCs) samples identified among anti-PLAR2 negative patients enrolled in the MONET study, who provided consent to store their samples collected during the follow-up at the Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica (BG).
  Interventions: Diagnostic Test: Flow-cytometry tetramer-based antigen-bait assay
- PBMCs isolated from volunteers (No Intervention): PBMCs isolated from volunteer subjects without a history of renal diseases, autoimmune disorders, diabetes mellitus, or current allergies, and who have undergone a one-week washout from antibiotics, anti-inflammatory medications, and antihistamines.

INTERVENTIONS:
Diagnostic Test: Flow-cytometry tetramer-based antigen-bait assay — For tetramer assembly, recombinant biotinylated PLA2R will be incubated with either streptavidin-PE (Agilent) or streptavidin-APC (Agilent) conjugates according to the NIH protocol (https://tetramer.yerkes.emory.edu/support/protocols#10).
  PBMCs will be thawed and resuspended in antibody cocktail medium containing 7.5ug APC- and PE- PLA2R tetramers. Multicolor flow cytometry will be used to identify B-cell subsets with standard technique and equipment (FACS FortessaX20, BD Biosciences and FlowJo software). PLA2R-specific B cells will be determined as Tetramer double (PE/APC) positive B cells that bind with proportional fluorescent intensities to each tetramer. Each sample will be incubated with only streptavidin-PE/APC conjugates to exclude B cells binding to the fluorochrome portion of the tetramers. T cell- and NK/NKT cell phenotyping will be assessed by FACS using ad-hoc antibody panels.
  Arms: PBMCs from MONET patients negative for anti-PLAR2; PBMCs from MONET patients positive for anti-PLAR2; PBMCs from ORION patients negative for anti-PLAR2; PBMCs from ORION patients positive for anti-PLAR2

SUMMARY:
This is a non-pharmacological interventional monocentric study to primarily assess the levels of circulating phospholipase A2 receptor (PLA2R)-specific B cells in patients with PLA2R-mediated MN enrolled in the ORION and MONET studies, before and at the different time points after therapy. It will also compare the phenotype of circulating PLA2R-specific B cell subsets over time in patients who achieved long-term remission, who experience MN relapses or did not respond to Obinutuzumab or Felzartamab therapies, and evaluate changes in lymphocyte subpopulations, including T cells and NK cells, possibly involved in the autoimmune process and in the response to B-cell depleting therapy.

DETAILED DESCRIPTION:
Primary Membranous Nephropathy (MN) is the most frequent cause of Nephrotic Syndrome (NS) in adults. Even though 30% of affected patients may experience spontaneous remission of the disease, MN-associated NS can severely impact on renal survival, with one third of patients invariably progressing to end-stage renal disease. In addition, NS, characterized clinically by massive proteinuria, hypoalbuminemia and generalized edema, severely affects patients' quality of life and may cause potentially life-threatening complications, including cardiovascular, thrombotic and infectious events.

MN is histologically characterized by the deposition of IgG4 and C3 on the subepithelial layer of the glomerular capillary wall, with variable degrees of glomerular basement membrane thickening. The discovery of autoantibodies directed against the M-type phospholipase A2 receptor (PLA2R) in 70% of patients finally proved MN as an autoimmune disease and provided the rationale for targeted therapies against the immune B-cell compartment.

The anti-CD20 chimeric monoclonal antibody Rituximab (RTX) is becoming the first-line therapy of MN treatment, being superior in inducing disease remission with lower incidence of adverse effects than generalized immunosuppression with glucocorticoids, alkylating agents or cyclosporine.

Binding of RTX to its molecular target results in a profound B-cell depletion in the peripheral blood, which persists for several months. In anti-PLA2R positive MN patients treated with RTX, B-cell depletion is frequently followed by a decrease in the autoantibody titer and by remission of the NS, suggesting that the drug may be active against the B-cell clones responsible for the production of anti-PLA2R antibodies.

However, the drug is effective only in 60% of cases, with the rest of patients remaining heavily proteinuric; in these patients anti-PLA2R antibodies persist after an initial transient decrease. In addition, approximately one third of patients that initially achieved clinical remission with RTX experience one or more disease relapses (usually associated with reappearance of autoantibodies), which might eventually become rituximab-dependent and spend most of their lives with nephrotic range proteinuria.

The reasons pertaining to the inter-individual differences in RTX efficacy, despite the evidence of a complete, homogenous peripheral blood B-cell depletion in all MN patients, are currently unknown.

Incomplete elimination of autoreactive B-cell clones in secondary lymphoid organs or persistence of long-lived autoantibody-producing cells in the bone marrow have been proposed as possible explanations for resistance to RTX treatment, but access to these compartments is technically difficult and phenotyping of peripheral B cells with conventional lineage markers may provide little information about the pathogenic process. Indeed, autoreactive B cells bearing a PLA2R-specific surface Ig receptor, as well as anti-PLA2R-producing PB/PC, are inevitably a very small fraction of the total circulating B-cell pool, and differences between groups may be easily missed if these subsets are not specifically accounted for. Consistent with this view, a recent study did not report any difference in B-cell subsets at baseline between MN patients who achieved remission after RTX infusion and RTX-resistant patients.

On the other hand, antibody-producing cells, i.e. plasmablasts (PB) and plasma cells (PC) do not express the CD20 molecule and are therefore not susceptible to RTX-induced lysis. In patient responding to RTX it could be possible that depletion of the B-cell pool (including antigen-experienced memory B cells) from which PB/PC originate may account for the effects of RTX on autoantibody levels, since a consistent fraction of these cells are short-lived.

- The ORION study (NCT05050214) The ORION study is a multicenter single-arm pilot clinical trial, designed to assess whether Obinutuzumab may safely achieve disease remission in Rituximab-Intolerant and Rituximab-Resistant patients with MN-associated nephrotic range proteinuria.

Obinutuzumab is a humanized, third-generation type II glycoengineered anti-CD20 monoclonal antibody which binds CD20 through a different orientation than rituximab and over a larger epitope. It appears to have more potent activity through Natural Killer (NK) cell-mediated antibody-dependent cellular cytotoxicity effect, enabling a more profound depletion of B lymphocytes - affecting even B lymphocytes in secondary lymphoid organs - as compared to rituximab.

ORION working hypothesis is that, in Rituximab-Resistant patients, RTX induced an incomplete B-cell depletion in secondary lymphoid organs due to CD20 internalization after antibody binding (i.e. antigenic modulation). This notion has been supported by several lines of evidence in other conditions, which showed persistence of B cells in primary and secondary lymphoid organs after high doses of rituximab despite complete depletion of these subsets from the circulation. Incomplete B-cell depletion may result in persistence of autoreactive memory B-cell clones that, upon proliferation and differentiation into antibody-secreting cells, could sustain disease activity and render the treatment ineffective. This may explain why in these patients, rituximab fails to reduce circulating autoantibodies and achieve disease remission, despite effective depletion of circulating B cells comparable to that observed in rituximab-sensitive patients. If the working hypothesis is correct, Obinutuzumab will achieve complete depletion of autoreactive B cells in these subjects, along with negativization of anti-PLA2R antibodies and remission of proteinuria.

ORION study has recently completed the 1-year follow-up of 20 patients with primary MN (17 rituximab-resistant and 3 rituximab-intolerant). During the follow-up peripheral blood mononuclear cells have been collected and stored in our lab facility.

- The MONET study (NCT04893096) The MONET study is an open-label, phase II study aimed at evaluating the effect of the anti-CD38 Antibody MOR202 (Felzartamab) in Patients with Membranous Nephropathy who Failed anti-CD20 target therapy.

MONET working hypothesis is that in patients with MN refractory to CD20-targeted therapy, the production of nephritogenic autoantibodies is sustained by mechanisms that do not depend on autoreactive CD20+ B cells. In such cases, autoantibodies could be produced by long-lived plasma cells that do not express the CD20 antigen on their surface, survive in bone marrow niches and do not depend on B-cell proliferation and differentiation. Indeed, in autoimmune diseases, long-lived autoreactive plasma cells largely resist B-cell targeted therapy, and these non-eradicated plasma cells continue to produce autoantibodies. Recently, it was shown that CD19-negative bone marrow plasma cells, which express CD38, are enriched in chronically inflamed tissue and secrete autoantibodies. Thus, while CD38-targeting antibodies were initially developed to target malignant plasma cells, these monoclonal antibodies may also abrogate the production of autoantibodies in autoimmune disorders and thereby reduce autoantibody-dependent effector mechanisms. Therefore, CD38-targeted therapy with MOR202 may abrogate autoantibody-dependent mechanisms in patients with plasma-cell mediated forms of MN who failed previous treatment with rituximab and second-generation anti-CD20 monoclonal antibodies such as ofatumumab.

MONET study has recently completed the 1-year follow-up of 9 patients with rituximab-resistant primary MN. During the follow-up, Peripheral Blood Mononuclear Cells (PBMCs) have been collected and stored in our lab facility.

- The PEPTIDE study (NCT04095156) The PEPTIDE study is aimed at analyzing the circulating immune repertoire of MN patients before and after the infusion of B cell depleting agents. As a complete novelty, circulating PLA2R-specific B cells are being assessed through a flow-cytometry-based antigen-bait assay.

The investigators recently set up and validated the methodology for the identification, enumeration and monitoring of B cells bearing a PLA2R-specific surface Ig using fluorochrome-labelled PLA2R tetramers built with recombinant monobiotinylated PLA2R protein and APC- and PE- streptavidin conjugated (manuscript in preparation).

Preliminary data from cohorts of RTX-resistant and -sensitive MN patients studied during the 12-month follow-up after therapy suggest that RTX failed to deplete PLA2R-specific B cells that persist following the anti-CD20 therapy in RTX-resistant MN patients. At variance, PLA2R-specific B cells significantly decreased post-treatment compared to baseline levels in patients achieving disease remission.

Based on all the above evidence, the investigators aim to apply the flow-cytometry-based antigen-bait assay methodology to monitor PLA2R-specific B cells in patients enrolled in ORION and MONET studies to get insight into the effect of Obinutuzumab and Felzartamab in MN patients in whom RTX failed to induce remission.

ELIGIBILITY:
Patients

Inclusion Criteria:

* Patients enrolled in the ORION and MONET studies who have who provided written informed consent to store their samples collected during the follow-up at the Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica (BG).

Exclusion Criteria:

* No written informed consent to store their samples collected during the follow-up at the Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica (BG).

Volunteers

Inclusion criteria:

* Adult males and females.
* Written informed consent.

Exclusion criteria:

* History of renal diseases, autoimmune disorders, diabetes mellitus, current allergies.
* Subjects who have taken antibiotics, anti-inflammatory drugs, or antihistamines within the past 7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Levels of circulating PLA2R-specific B cells | Levels measured at baseline and at 3, 6, 9, 12, 18, 24 months.
  Levels of circulating PLA2R-specific B cells in patients with PLA2R-mediated MN enrolled in the ORION study
Levels of circulating PLA2R-specific B cells | Levels measured at baseline, 29, 141 days and at 6, 9, 12, 18, 24 months.
  Levels of circulating PLA2R-specific B cells in patients with PLA2R-mediated MN enrolled in the MONET studies

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, M.D., Study Director — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- Clinical Research Centre for Rare Diseases Aldo e Cele Daccò, Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruggenenti P, Debiec H, Ruggiero B, Chianca A, Pelle T, Gaspari F, Suardi F, Gagliardini E, Orisio S, Benigni A, Ronco P, Remuzzi G. Anti-Phospholipase A2 Receptor Antibody Titer Predicts Post-Rituximab Outcome of Membranous Nephropathy. J Am Soc Nephrol. 2015 Oct;26(10):2545-58. doi: 10.1681/ASN.2014070640. Epub 2015 Mar 24. PMID 25804280
- [Background] Beck LH Jr, Fervenza FC, Beck DM, Bonegio RG, Malik FA, Erickson SB, Cosio FG, Cattran DC, Salant DJ. Rituximab-induced depletion of anti-PLA2R autoantibodies predicts response in membranous nephropathy. J Am Soc Nephrol. 2011 Aug;22(8):1543-50. doi: 10.1681/ASN.2010111125. Epub 2011 Jul 22. PMID 21784898
- [Background] Beck LH Jr, Bonegio RG, Lambeau G, Beck DM, Powell DW, Cummins TD, Klein JB, Salant DJ. M-type phospholipase A2 receptor as target antigen in idiopathic membranous nephropathy. N Engl J Med. 2009 Jul 2;361(1):11-21. doi: 10.1056/NEJMoa0810457. PMID 19571279